CLINICAL TRIAL: NCT01996098
Title: A Multicenter, Randomized, Phase III Trial of Chemotherapy Followed by 6-month or 12-month Icotinib Versus Chemotherapy as Adjuvant Therapy in Stage IIA-IIIA Non-small Cell Lung Cancer Harboring Epidermal Growth Factor Receptor Mutation
Brief Title: Icotinib Following Chemotherapy Versus Chemotherapy as Adjuvant Therapy in Stage IIA-IIIA NSCLC With EGFR Mutation
Acronym: ICTAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accural.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1002; wsy003 (Other: Guangdong Province Association Study of Thoracic Oncology)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 6-month icotinib (Experimental): Icotinib 125 mg three times daily (375 mg per day) by mouth for 6 months
  Interventions: Drug: 6-month Icotinib
- 12-month icotinib (Experimental): Icotinib 125 mg three times daily (375 mg per day) by mouth for 12 months
  Interventions: Drug: 12-month icotinib
- Chemotherapy alone (No Intervention): No intervention

INTERVENTIONS:
Drug: 6-month Icotinib — 125 mg three times daily (375 mg per day) by mouth for 6 months
  Other Names: BPI-2009; Conmana
  Arms: 6-month icotinib
Drug: 12-month icotinib — 125 mg three times daily (375 mg per day) by mouth for 12 months
  Other Names: BPI-2009; Conmana
  Arms: 12-month icotinib

SUMMARY:
The purpose of this study is studying icotinib following chemotherapy to see how well it works compared to chemotherapy in treating patients with resected stage IIA-IIIA NSCLC harboring EGFR mutation.

DETAILED DESCRIPTION:
Adjuvant chemotherapy is recommended for routine use in patients with fully resected stage IIA-IIIA non-small cell lung cancer (NSCLC). Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) show great efficacy in patients with advanced non-small cell lung cancer (NSCLC) with EGFR mutation. Icotinib is a novel EGFR-TKI developed by a group of Chinese scientists. In the phase III ICOGEN trial, icotinib had non-inferiority efficacy to gefitinib with better safety. In phase II trial, chemotherapy followed by 6-month gefitinib as adjuvant therapy can confer longer disease-free survival compared with chemotherapy alone in patients with resected stage IIIA-N2 non-small cell lung cancer harboring EGFR mutations. This study is to studying 6-month or 12-month icotinib following chemotherapy to see how well it works compared to chemotherapy in treating patients with resected stage IIA-IIIA NSCLC harboring EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Aged 18-75 years.
* Had completely resected pathological confirmed stage IIA-IIIA NSCLC.
* EGFR activating mutation in exon 19 or 21.
* Had completed four cycles of platinum-based adjuvant chemotherapy.
* Able to start the investigational therapy within 4 weeks after the completion of four cycles of adjuvant chemotherapy.
* ECOG performance status of 0-1.
* Had a life expectancy of 12 weeks or more.
* Adequate hematological function, adequate liver function and renal function.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Female patients, except those who are postmenopausal or surgically sterilized, must have a negative pre-study serum or urine pregnancy test.

Exclusion Criteria:

* Had had previous chemotherapy besides four cycles of adjuvant chemotherapy, radiotherapy, or agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Had a history another malignancy in the last 5 years with the exception of cured basal cell carcinoma of the skin, cured in situ carcinoma of the uterine cervix and cured epithelial carcinoma of the bladder.
* Any evidence confirmed tumor recurrence before investigational therapy.
* Known severe hypersensitivity to icotinib or any of the excipients of this product.
* Evidence of clinically active interstitial lung disease.
* Eye inflammation not fully controlled or conditions predisposing the subject to this.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Known human immunodeficiency virus (HIV) infection.
* Pregnancy or breast-feeding women.
* Ingredients mixed with small cell lung cancer patients.
* History of neurologic or psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival | 5 years after the last patient is randomized
  Disease-free survival was assessed from randomization to disease recurrence or death as a result of any cause.

SECONDARY OUTCOMES:
Overall Survival | 5 years after the last patient is randomized
  Overall survival was assessed from randomization to death as a result of any cause.
Number of Participants with Adverse Events | 2 years
  To assess if the addition of icotinib to chemotherapy is safe.
Change from baseline in patient reported Lung Cancer Functional Assessment | 2 years
  Quality of life as measured by the Functional Assessment of Cancer Therapy - Lung Cancer (FACT-L) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China